CLINICAL TRIAL: NCT01030731
Title: An Open-Label Pharmacokinetic Study of Ceftobiprole in Healthy Volunteers and Patients With End Stage Renal Disease Receiving Hemodialysis
Brief Title: Pharmacokinetic Study,Ceftobiprole,Healthy Volunteers,Healthy Patients With End Stage Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR012448
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Staphylococcal Skin Infections; Streptococcal Infections
Keywords: Renal Dialysis, Ceftobiprole; Skin and soft tissue Infections; Staphylococcal Skin Infections; Streptococcal Infection
MeSH Terms: conditions — Staphylococcal Skin Infections; Streptococcal Infections; Soft Tissue Infections | interventions — ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftobiprole (end-stage renal disease subjects). (Experimental): Ceftobiprole 250mg single dose over 2 hours.
  Interventions: Drug: Ceftobiprole
- Ceftobiprole (healthy subjects) (Active Comparator): Ceftobiprole 250 mg single dose over 2 hours.
  Interventions: Drug: Ceftobiprole

INTERVENTIONS:
Drug: Ceftobiprole — Ceftobiprole 250mg single dose over 2 hours.

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) of ceftobiprole after a single 250-mg intravenous (IV) infusion (given directly into the vein) for 2 hours, before and after dialysis to patients with end-stage renal disease (ESRD) requiring hemodialysis or healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) of ceftobiprole after a single 250-mg intravenous (IV) infusion (given directly into the vein) for 2 hours, before and after dialysis to patients with end-stage renal disease (ESRD) requiring hemodialysis or healthy volunteers. This is a Phase 1, open label study (all patients involved know the identity of the drug). Healthy volunteers will be given a single 2-hour infusion of 250 mg ceftobiprole; patients with ESRD on hemodialysis will be given a 2-hour infusion of 250 mg ceftobiprole 3 hours either before dialysis or immediately after dialysis. Plasma and urine samples will be assayed for ceftobiprole. Samples will be collected over a 48 hour period of time. Safety evaluations will include monitoring of adverse events, clinical laboratory tests (hematology and serum chemistry in all patients/volunteers, and urinalysis in healthy volunteers subjects), pregnancy testing, vital signs, physical examination, and recording of concomitant medications. Healthy volunteers will be given a single 2-hour infusion of 250 mg ceftobiprole; patients with ESRD on hemodialysis will be given a 2-hour infusion of 250 mg ceftobiprole 3 hours either before dialysis or immediately after dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer or be a hemodialysis patient in stable physical condition with a diagnosis of ESRD and requiring hemodialysis treatment 3 times per week

Exclusion Criteria:

* History of repeated severe nausea
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Recent febrile illness

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of ceftobiprole and its open-ring metabolite in patients undergoing dialysis. | Days 1 through 3 of study period 1 for healthy volunteers with normal renal function and Days 1 through 5 of study period 1 (predialysis) and study period 2 (postdialysis) for patients with ESRD

SECONDARY OUTCOMES:
To assess the safety and tolerability of ceftobiprole in patients with ESRD undergoing dialysis and in a control group of healthy volunteers with normal renal function | 31 days for healthy volunteers and 52 days for patients with ESRD, including the screening, treatment, end-of-study, and follow-up phase
To compare the pharmacokinetics of ceftobiprole and its open-ring metabolite in patients with ESRD undergoing hemodialysis with a control group of healthy volunteers with normal renal function | Days 1 through 3 of study period 1 for healthy volunteers with normal renal function and Days 1 through 5 of study period 1 (predialysis) and study period 2 (postdialysis) for patients with ESRD
To determine the extent of the ceftobiprole dose removed by hemodialysis | Days 1 through 3 of study period 1 for healthy volunteers with normal renal function and Days 1 through 5 of study period 1 (predialysis) and study period 2 (postdialysis) for patients with ESRD

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Pharmacokinetic Study of Ceftobiprole in Healthy Volunteers and Patients With End Stage Renal Disease Receiving Hemodialysis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=746&filename=CR012448_CSR.pdf